CLINICAL TRIAL: NCT00005821
Title: Sentinel Lymph Node Biopsy in the Assessment of Axillary Nodal Status in Operable Breast Cancer
Brief Title: Sentinel Lymph Node Biopsy to Assess Axillary Lymph Nodes in Women With Stage I or Stage II Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067828; RMNHS-1631; EU-20006
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2003-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — iso-sulfan blue; Sentinel Lymph Node Biopsy

INTERVENTIONS:
Drug: patent blue V dye
Procedure: conventional surgery
Procedure: lymphangiography
Procedure: radionuclide imaging
Procedure: sentinel lymph node biopsy
Radiation: Technetium Tc 99m human serum albumin colloid

SUMMARY:
RATIONALE: Diagnostic procedures such as sentinel lymph node biopsy may improve the ability to detect breast cancer and determine the extent of disease.

PURPOSE: Phase II trial to study the effectiveness of sentinel lymph node biopsy to assess axillary lymph nodes in women who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare sentinel node biopsy vs axillary dissection in determining axillary nodal status in women with resectable stage I or II breast cancer.

OUTLINE: Patients are stratified according to node status (positive vs negative).

Patients undergo lymphoscintigraphy, which consists of technetium Tc 99m human serum albumin colloid being injected near the tumor. Dynamic imaging using a gamma camera is performed for 20 minutes postinjection and static images are obtained for up to 3 hours postinjection.

Surgery is performed within 24 hours of lymphoscintigraphy. Patients are injected with patent blue V dye near the tumor and a gamma detection probe is used to measure radioactive counts in the sentinel node. Surgery begins within 5 minutes of the patent blue V dye injection.

All lymph nodes that stain blue or have a high radioactive count are removed. The primary breast lump is removed by either wide local excision or mastectomy and the axilla are cleared by standard axillary dissection.

Some patients may only receive patent blue V dye injected as a pilot study. Sentinel lymph node biopsy and axillary dissection proceed as above.

PROJECTED ACCRUAL: A total of 150 patients (75 per stratum) will be accrued for the main study plus another 50 patients for the pilot study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I or II invasive breast cancer by triple assessment:

  * Clinically
  * Mammogram and/or ultrasound
  * Fine needle cytology
* Resectable disease by either wide local excision or mastectomy with axillary dissection
* No ductal carcinoma in situ
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant
* No known allergy to vital blue dye
* No mental illness or handicap that would preclude study entry
* No other severe illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gui, MD, MS, FRCS(Edin), FRCS(Eng), Study Chair — Royal Marsden NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - St. George's Hospital, London, England
  - Royal Marsden NHS Trust, London, England
  - Royal Brompton National, Heart and Lung Hospital, London, England
  - Royal Marsden Hospital, Sutton, England